CLINICAL TRIAL: NCT04610567
Title: Two Phases Clinical Trial to Evaluate Safety and Efficacy of Methotrexate Associated to LDL Like Nanoparticles (LDE-MTX) in the Treatment of Patients With Mild Coronavirus-19 (COVID-19) Disease.
Brief Title: Treatment of Patients With Mild Coronavirus-19 (COVID-19) Disease With Methotrexate Associated to LDL Like Nanoparticles (Nano-COVID19)
Acronym: Nano-COVID19
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Hospital Santa Marcelina (Other)
Responsible Party: Principal Investigator, Raul Cavalcante Maranhão, MD; PHD. Director Lipid Metabolism Laboratory, Heart Institute, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 36746020.5.1001.0068
Record Dates: First submitted 2020-10-24; First posted 2020-10-30 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Coronavirus; Inflammation; Covid19
Keywords: coronavirus; inflammation; nanoparticles; methotrexate; covid19
MeSH Terms: conditions — Coronavirus Infections; Inflammation; COVID-19

STUDY DESIGN:
Intervention Model Description: This will be a randomized, double-blind, placebo-controlled, multi-center study.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- MTX-LDE phase 1 (Experimental): Methotrexate carried by a lipid nanoparticle (MTX-LDE)
  Interventions: Drug: Methotrexate-LDE phase 1
- MTX-LDE phase 2 (Experimental): Methotrexate carried by a lipid nanoparticle (MTX-LDE)
  Interventions: Drug: Methotrexate-LDE phase 2
- Placebo-LDE phase 2 (Placebo Comparator): Lipid nanoparticle (LDE)
  Interventions: Drug: Placebo-LDE phase 2

INTERVENTIONS:
Drug: Methotrexate-LDE phase 1 — 3 patients will receive MTX-LDE at the dose of 15mg IV each 7 days during hospitalization, up to 3 times . After that, 9 patients will receive MTX-LDE at the dose of 30mg IV each 7 days during hospitalization, up to 3 times .
  All patients will receive Leucovorin (calcium foliate) 25mg IV, 24hr after administration of MTX-LDE
  Other Names: MTX-LDE phase 1
  Arms: MTX-LDE phase 1
Drug: Methotrexate-LDE phase 2 — 44 patients will receive MTX-LDE at the dose of 30mg IV each 7 days during hospitalization, up to 3 times dose of 30mg IV each 7 days during hospitalization, up to 3 times . All patients will receive Leucovorin (calcium foliate) 25mg IV, 24hr after administration of MTX-LDE
  Other Names: MTX-LDE phase 2
  Arms: MTX-LDE phase 2
Drug: Placebo-LDE phase 2 — 44 patients will receive Placebo-LDE IV each 7 days during hospitalization, up to 3 times dose of 30mg IV each 7 days during hospitalization, up to 3 times . All patients will receive Leucovorin (calcium foliate) 25mg IV, 24hr after administration of Placebo-LDE
  Arms: Placebo-LDE phase 2

SUMMARY:
The investigators propose a prospective, randomized, double-blind, placebo-controlled study, conducted in two phases. The purpose of the study is to evaluate the safety and efficacy of methotrexate in a cholesterol-rich non-protein nanoparticle (MTX -LDE) in adults diagnosed with mild Coronavirus-19(COVID-19) disease.

A total of 100 patients will be randomized to receive MTX-LDE or placebo each 7 days, up to 3 times, during in hospital treatment.

DETAILED DESCRIPTION:
The objective of the study is to evaluate the safety and efficacy of (MTX -LDE) in patients with mild Coronavirus-19 (COVID-19) disease.

In phase 1, firstly 3 patients with moderate COVID-19 disease will receive MTX-LDE IV 15mg each 7 days, up to 3 times, during hospitalization. After that, 9 patients with moderate COVID-19 disease will receive MTX-LDE IV 30mg each 7 days, up to 3 times, during hospitalization. Follow-up assessments will occur daily following randomization during in hospital treatment and 2 weeks after discharge for evaluation of the occurrence of adverse events.The purpose of this phase will be evaluate safety and pharmacokinetics.

If no objection by data and safety monitoring board (DSMB), will be authorized to start the second phase.

In phase 2, 88 patients with moderate COVID-19 disease will be randomized to receive MTX-LDE IV 30mg or placebo-LDE IV each 7 days, up to 3 times, during hospitalization. Follow-up assessments will occur daily following randomization during in hospital treatment and 2 weeks after discharge for evaluation of the occurrence of any trial endpoints or other adverse events.The primary endpoint of this phase will be reduction in duration of hospitalization stay between groups.

Patients will undergo clinical and laboratory safety evaluations daily. An algorithm for drug suspension based on clinical and laboratory finding will be followed.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were hospitalized with confirmed COVID-19
* Mild Coronavirus-19 disease (WHO Coronavirus-19 scale < 5)
* Fewer than 14 days since symptom onset.
* Female patient is not of childbearing potential, defined as postmenopausal for at least 1 year or surgically sterile.
* Female patient is of childbearing potential must has a negative pregnancy test.
* Signing the study informed consent.

Exclusion Criteria:

* Need for oxygen supplementation >4 L/min via nasal cannula or ≥40% via Venturi mask.
* Need for oxygen supplementation via high-flow nasal cannula.
* Need for invasive mechanical ventilation.
* Extent of pulmonary involvement > 50% by CT scan.
* Chronic renal failure (estimated glomerular filtration rate <30 mL/min/1.73 m2)
* History of liver cirrhosis (Bilirubins levels > 3mg/dl)
* History of heart failure ( Ejection fraction <40%)
* History of Steven-Johnson disease
* History of stroke in the last 6 months
* History of sickle cell disease
* Chronic use of oral steroid therapy or other immunosuppressive or biologic response modifiers.
* Prior history of chronic hepatitis B or C infection and known HIV positive.
* Patient undergoing chemotherapy for cancer
* Sepsis caused by fungal or multidrug resistant gram-negative bacteria
* Known allergy to methotrexate.
* Body mass index(BMI) > 40 or <18.5
* Pregnancy or breastfeeding.
* Patients enrolled in other clinical trials in the last 12 months
* Patient is considered by the investigator, for any reason, to be an unsuitable candidate for the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-10-27 (Actual); Primary Completion 2021-03-15 (Estimated); Study Completion 2021-07-15 (Estimated)

PRIMARY OUTCOMES:
Duration of hospital stay | 30 days after randomization
  Compare the duration of hospital stay between groups

SECONDARY OUTCOMES:
Number of participants requiring mechanical ventilation | 15 days after randomization
  The secondary outcome is the need for mechanical ventilation between groups
Number of participants requiring vasoactive drugs | 15 days after randomization
  The secondary outcome is the need for vasoactive drugs between groups
Number of participants requiring renal replacement therapy | 15 days after randomization
  The secondary outcome is the need for renal replacement therapy between groups
Incidence of secondary infection | 15 days after randomization
  The secondary outcome is the incidence of secondary infection between groups
Sequential Organ Failure Assessment (SOFA) score | Baseline and change from baseline to 15 days after randomization
  The secondary outcome is the comparison of Sequential Organ Failure Assessment (SOFA) score between groups
World Health Organization (WHO) COVID-19 score | Baseline and change from baseline to 15 days after randomization
  The secondary outcome is the comparison of World Health Organization (WHO) COVID-19 clinical score between groups
Interleukin 6 (IL-6) | Baseline and change from baseline to 15 days after randomization
  The secondary outcome is the comparison of IL-6 levels between groups
Dimer-D | Baseline and change from baseline to 15 days after randomization
  The secondary outcome is the comparison of dimer-D levels between groups
Chest CT scan | Baseline and change from baseline to 15 days after randomization
  The secondary outcome is the comparison of chest CT scan between groups
Incidence and severity of laboratory alterations | 30 days after randomization
  The secondary outcome is the comparison of red blood cells; white blood cells;Platelets; Urea;Creatinine levels between groups
Clinical side effects | 30 days after randomization
  Compare the incidence of clinical significant symptoms (new and persistent stomatitis, vomiting, diarrhea, alopecia, neurotoxicity, bradycardia, hypotension, local pain) reported between groups.
Other adverse events | 30 days after randomization
  Compare the incidence of other adverse events (not expected) between groups

CONTACTS AND LOCATIONS:
Locations (3):
- Brazil (3):
  - Heart Institute (InCor) - University of São Paulo Medical School, São Paulo, Brazil, São Paulo, São Paulo
  - Hospital Santa Marcelina, São Paulo, São Paulo
  - Institute Prevent Senior, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu PP, Blet A, Smyth D, Li H. The Science Underlying COVID-19: Implications for the Cardiovascular System. Circulation. 2020 Jul 7;142(1):68-78. doi: 10.1161/CIRCULATIONAHA.120.047549. Epub 2020 Apr 15. PMID 32293910
- [Background] Solinas C, Perra L, Aiello M, Migliori E, Petrosillo N. A critical evaluation of glucocorticoids in the management of severe COVID-19. Cytokine Growth Factor Rev. 2020 Aug;54:8-23. doi: 10.1016/j.cytogfr.2020.06.012. Epub 2020 Jun 24. PMID 32616381
- [Background] Vinciguerra M, Romiti S, Fattouch K, De Bellis A, Greco E. Atherosclerosis as Pathogenetic Substrate for Sars-Cov2 Cytokine Storm. J Clin Med. 2020 Jul 3;9(7):2095. doi: 10.3390/jcm9072095. PMID 32635302
- [Background] Zhang S, Li L, Shen A, Chen Y, Qi Z. Rational Use of Tocilizumab in the Treatment of Novel Coronavirus Pneumonia. Clin Drug Investig. 2020 Jun;40(6):511-518. doi: 10.1007/s40261-020-00917-3. PMID 32337664
- [Background] Barbieri LR, Lourenco-Filho DD, Tavares ER, Carvalho PO, Gutierrez PS, Maranhao RC, Stolf NAG. Influence of Drugs Carried in Lipid Nanoparticles in Coronary Disease of Rabbit Transplanted Heart. Ann Thorac Surg. 2017 Aug;104(2):577-583. doi: 10.1016/j.athoracsur.2016.12.044. Epub 2017 Mar 24. PMID 28347533
- [Background] Bulgarelli A, Leite AC Jr, Dias AA, Maranhao RC. Anti-atherogenic effects of methotrexate carried by a lipid nanoemulsion that binds to LDL receptors in cholesterol-fed rabbits. Cardiovasc Drugs Ther. 2013 Dec;27(6):531-9. doi: 10.1007/s10557-013-6488-3. PMID 24065615
- [Background] Bulgarelli A, Martins Dias AA, Caramelli B, Maranhao RC. Treatment with methotrexate inhibits atherogenesis in cholesterol-fed rabbits. J Cardiovasc Pharmacol. 2012 Apr;59(4):308-14. doi: 10.1097/FJC.0b013e318241c385. PMID 22113347
- [Background] Maranhao RC, Tavares ER. Advances in non-invasive drug delivery for atherosclerotic heart disease. Expert Opin Drug Deliv. 2015 Jul;12(7):1135-47. doi: 10.1517/17425247.2015.999663. Epub 2015 Jan 14. PMID 25585820
- [Background] Maranhao RC, Guido MC, de Lima AD, Tavares ER, Marques AF, Tavares de Melo MD, Nicolau JC, Salemi VM, Kalil-Filho R. Methotrexate carried in lipid core nanoparticles reduces myocardial infarction size and improves cardiac function in rats. Int J Nanomedicine. 2017 May 17;12:3767-3784. doi: 10.2147/IJN.S129324. eCollection 2017. PMID 28553113
- [Result] Shah A, Kashyap R, Tosh P, Sampathkumar P, O'Horo JC. Guide to Understanding the 2019 Novel Coronavirus. Mayo Clin Proc. 2020 Apr;95(4):646-652. doi: 10.1016/j.mayocp.2020.02.003. Epub 2020 Feb 28. No abstract available. PMID 32122636
- [Result] Chen N, Zhou M, Dong X, Qu J, Gong F, Han Y, Qiu Y, Wang J, Liu Y, Wei Y, Xia J, Yu T, Zhang X, Zhang L. Epidemiological and clinical characteristics of 99 cases of 2019 novel coronavirus pneumonia in Wuhan, China: a descriptive study. Lancet. 2020 Feb 15;395(10223):507-513. doi: 10.1016/S0140-6736(20)30211-7. Epub 2020 Jan 30. PMID 32007143
- [Result] Mitchell WB. Thromboinflammation in COVID-19 acute lung injury. Paediatr Respir Rev. 2020 Sep;35:20-24. doi: 10.1016/j.prrv.2020.06.004. Epub 2020 Jun 11. PMID 32653469
- [Result] Zhou Z, Guo D, Li C, Fang Z, Chen L, Yang R, Li X, Zeng W. Coronavirus disease 2019: initial chest CT findings. Eur Radiol. 2020 Aug;30(8):4398-4406. doi: 10.1007/s00330-020-06816-7. Epub 2020 Mar 24. PMID 32211963
- [Result] Cronstein BN. Molecular therapeutics. Methotrexate and its mechanism of action. Arthritis Rheum. 1996 Dec;39(12):1951-60. doi: 10.1002/art.1780391203. No abstract available. PMID 8961899
- See also: WHO COVID-19 Therapeutic Trial Synopsis — https://www.who.int/docs/default-source/blue-print/covid-19-therapeutic-trial-synopsis.pdf?sfvrsn=44b83344_1&download=true.